CLINICAL TRIAL: NCT05955976
Title: Study to Compare the Characteristics of Hoffa Adipose Tissue and Intramuscular Adipose Tissue in the Quadriceps Muscle
Brief Title: Characteristics of Hoffa Adipose Tissue and Intramuscular Adipose Tissue in the Quadriceps Muscle
Acronym: ADIPENIGME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Rhumato02
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hoffa tissue (1 cm x 1 cm) and intramuscular fat tissue (1 cm x 1 cm)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suffering of knee ostheoarthritis undergoing a surgery for a total knee prosthesis.
  Interventions: Other: BIOPSY

INTERVENTIONS:
Other: BIOPSY — biopsy

SUMMARY:
Over the last few years, it has been suggested that Knee Ostheoarthritis (KOA) incidence and progression could potentially be related to skeletal muscle characteristics. In particular, weakness of the quadriceps muscle would be a key determinant of KOA. However the mechanisms underpinning the influence of skeletal muscle in the pathophysiology of ostheoarthritis (OA) are poorly understood.

Crosstalk between skeletal muscle and structures around and in the joint is of interest. In physical deconditioning and aging, it has been reported that skeletal muscle can be replaced by adipose tissue. Several factors involved in the development of OA but also of adipose tissue may be involved in these muscular changes. Of interest, in patients with KOA, quadriceps weakness is an ubiquitous clinical finding. Infiltration of adipose tissue in skeletal muscle has been shown to affect muscle strength and mobility and be linked to cartilage volume loss and the occurrence/progression of KOA.

The main objective of this study is to compare the characteristics of the Hoffa tissus and the intamuscular fat (IMF) tissus in the quadriceps muscle in patients with gonarthrosis requiring total knee prosthesis.

This is a single-centre study based on a collection of surgical waste and is categorized as Research Not Involving Human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, aged between 40 and 85 years
* Patient having a confirmed diagnosis of knee ostheoarthritis
* Patient undergoing a surgery for a total knee prosthesis for knee ostheoarthritis

Exclusion Criteria:

-

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 40 and 85 years that have a scheduled surgery for a total knee prosthesis and have a confirmed diagnosis of knee ostheoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Comparison between Hoffa tissue and intramuscular fat tissue (quadriceps): adipose tissue size differences | 4 months
  size mesured in mm
Comparison between Hoffa tissue and intramuscular fat tissue (quadriceps): lipid levels | 4 months
  level mesured in %
Comparison between Hoffa tissue and intramuscular fat tissue (quadriceps):fibrotic tissue | 4 months
  rate mesured in %

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France